CLINICAL TRIAL: NCT05397704
Title: Cyban Brain Pulse Oximeter Study
Brief Title: Brain Oximeter Calibration and Validation Study
Acronym: TPOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyban Pty Ltd (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00110458
Record Dates: First submitted 2022-05-24; First posted 2022-05-31 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Brain Injuries, Traumatic
Keywords: hypoxia
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypoxia

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- desaturation (Experimental): Controlled desaturation studies are conducted by changing the alveolar oxygen tension (or pressure, PAO2). This is achieved by a dedicated gas delivery system, RespirAct RAMR (Thornhill Research, Toronto, ON). The attained PAO2 then determines the arterial oxygen tension (PaO2) at the alveolar-arterial interspace in the lung. The arterial oxygen tension (PaO2) will then determine the arterial oxygen saturation (SaO2) and in turn, the pulse oximeter oxygen saturation (SpO2). The step down changes in the alveolar oxygen tension (PAO2) will result in the corresponding step down changes in SaO2/SpO2 from 100 to 70%.
  Interventions: Device: brain pulse oximeter

INTERVENTIONS:
Device: brain pulse oximeter — brain oxygen monitoring during hypoxia

SUMMARY:
The purpose of the study is to calibrate and to validate the accuracy of the oximeter with an estimate of brain oxygen levels assessed by measuring arterial and internal jugular vein blood oxygen saturations.

DETAILED DESCRIPTION:
The device is a non invasive NIRS monitor. It detects signals from which are derived venous and arterial blood brain oxygen levels.

The device will be used as a adjunct monitor in patients with a brain injury or at risk of a brain injury.

The primary objective of the study is to measure the absolute and relative accuracy of the StO2 device by comparing the NIRS-derived brain tissue oxygen saturation with blood-referenced CO-oximeter oxygen saturation values. The CO-oximeter oxygen saturation values from paired arterial and internal jugular venous blood gas samples are then inserted into a weighted-equation to derive the calculated brain tissue oxygen saturation. Accuracy is reported over a range of oxygen saturations with study subjects exposed to a controlled oxygen desaturation with serial sampling of paired arterial and internal jugular venous blood gas samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female subjects between the ages of 18 to 45 years;
* Completion of a health screening for a medical history by a licensed physician, nurse practitioner, or physician assistant;
* Minimum weight 40kg;
* BMI within range 18.0 - 35.0;
* Assigned American Society of Anesthesiologists (ASA) Physical Status 1 by Principal Investigator or delegate

Exclusion Criteria:

* Prior or known allergies to lidocaine (or similar pharmacologic agents, e.g., Novocain) [self- reported];
* Prior known severe allergies to medical grade adhesive/tape (Band-Aid) [self-reported];
* Taking any medication other than birth control[self-reported];
* Is currently participating in, or has recently participated in (discontinued within 30 days prior to the hypoxia procedure for this study) in an investigational drug, device, or biologic study [self- reported];
* Has a negative Allen's Test to confirm non- patency of the collateral artery [clinical assessment by PI or delegate];
* Has made a whole blood donation or has had at least 450 ml of blood drawn within 8 weeks prior to the study procedure [self-reported];
* Is female with a positive pregnancy test [serum or urine], or is female and is unwilling to use effective birth control between the time of screening and study procedure or is breast feeding;
* Has anemia [lab values specific for gender];
* Has heparin allergy
* Has a history of sickle cell trait or thalassemia [self-reported];
* Has an abnormal hemoglobin electrophoresis result [lab measurement];
* Has a positive urine cotinine test or urine drug screen or oral ethanol test;
* Has a room air saturation less than 95% by pulse oximetry [measurement by PI or delegate]
* Has a clinically significant abnormal EKG [assessment by PI or delegate];
* Has a clinically significant abnormal pulmonary function test via spirometry [assessment by PI or delegate];
* Has a COHb greater than 3%, or MetHb greater than 2% [measured by venous blood sample co- oximetry].

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of brain pulse oximeter | Data will be collected over a 90 minute period for each patient
  Bland Altman analysis

CONTACTS AND LOCATIONS:
Overall Officials: David MacLeod, MBBS, Principal Investigator — Duke University
Locations (1):
- Duke Hospital Human Pharmacology & Physiology Lab, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No